CLINICAL TRIAL: NCT06662136
Title: The Effect of Health Belief Model-Based Motivational Interviews on Women's HPV-DNA Testing According to the Precautionary Acceptance Process
Brief Title: The Effect of Motivational Interviewing on HPV-DNA Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muazez küçükkaya (Other)
Responsible Party: Sponsor-Investigator, Muazez küçükkaya, Principal Investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IstanbulUC-SBF-MK-1
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancers
Keywords: Human papillomavirus; Woman; Midwife
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: motivational interviewing to the experimental group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Participants in the experimental group will be given motivational interviews about HPV at 4 different times and will also be given an educational brochure.
  Interventions: Behavioral: motivasional intereview
- control group (No Intervention): Participants in the control group will not receive any intervention

INTERVENTIONS:
Behavioral: motivasional intereview — No application will be made to the participants in the control group
  Arms: Experimental group

SUMMARY:
The aim of this randomized controlled study was to examine the effects of Health Belief Model Based Motivational Interviewing on HPV-DNA testing in women according to the Precautionary Acceptance Process.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) infection is the main determinant of cervical cancer in women. Current studies indicate that cervical cancers are caused by sexually transmitted HPV infection and 84% of HPV-associated cancer lesions are cervical cancer. HPV infection causes more than 14 million people to become infected with HPV annually and 80% of sexually active individuals to become infected with HPV during their lifetime. Today, more than 200 HPV types have been identified. According to the International Agency for Research on Cancer, high-risk HPV genotypes including 16, 18, 31, 33, 45, 52, and 58 are responsible for approximately 90% of anogenital HPV-positive cancers worldwide, while low-risk genotypes HPV 6 and 11 are responsible for 90% of genital warts. Cancer is an important public health problem that increases the risk of mortality and morbidity in women all over the world. Gynecological cancers can be prevented by changing/abandoning risk factors, cases can be detected at an early stage with early diagnosis and screening programs, and a chance for treatment can be found. However, it is known that women do not apply to health institutions or postpone them due to reasons such as ignoring health problems, lack of information, embarrassment, and economic problems. The World Health Organization (WHO) emphasizes that at least one-third of cancer cases can be prevented with preventive care strategies and recommends the implementation of low-cost and long-term strategies in cancer control. All health professionals have important roles and responsibilities in the care and treatment processes in the successful implementation of cancer prevention, early diagnosis and screening programs. High cancer screening rates in the general population are associated with the health beliefs of the individual. According to the Health Belief Model (HBM); perceived barriers are the perceptions of factors that prevent or make it difficult to perform a protective behavior related to health. If individuals are sensitive that a health problem will seriously harm them, they think that the harm that will come to them will decrease when they take action. They believe that if they do not take action, more severe consequences may arise than the burden (cost, time, etc.) of the factors that create the perception of barriers. Motivational interviewing (MI) is a collaborative conversation style to strengthen a person's own motivation and commitment to change. Motivational interviewing is an evidence-based, successful intervention approach to facilitate positive behavioral change and is frequently used in substance abuse, mental health, primary and special health areas. Studies have shown the effectiveness of motivational interviews, especially SIM-based motivational interviews. The Precautionary Acceptance Process Model (PAPM) is a method that states that people may be in different motivational stages during the process of showing a behavior, therefore the same intervention applied to people evaluated in a single pot may not be effective for everyone, and the Precautionary Acceptance Process Model (PAPM), which is known to a limited extent in our country, is a suitable model especially in preventive health service practices, health protection and development programs. In the prevention of cervical cancer, health personnel working especially in primary health care services actively play a role in increasing the awareness levels of women in the society they serve and in directing them to early diagnosis. In this context, it is thought that midwives, especially those in the first stage, should be at the forefront with their education and consultancy roles in addition to their practitioner roles, as they reach women of all ages .

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-45 registered at Family Health Centre No. 1,
* Who currently have or have had an active sex life,
* Women who have not undergone an HPV-DNA test in the last five years,
* Women who can read and write, have no communication problems, and can use a smartphone and WhatsApp,
* Women with no diagnosed psychiatric problems,
* Women who agreed to participate in the study.

Exclusion Criteria:

* Women who were unable to complete the entire study due to any circumstances during the data collection phases,
* Women who voluntarily withdrew from the study were excluded.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Learning about HPV | From the beginning of the study until the 4th month.
  The program was planned as 4 sessions and the duration of the interview was 20-30 minutes. The women in the experimental group will be given 4 motivational interviews and a training brochure. Questionnaire/scale forms will be administered 4 times in total: The scales will be administered as a pre-test before the intervention, an interim test after the second motivational interview, a final test after the fourth motivational interview, and a final test two months after the last interview. The total score to be obtained from HPV-BÖ is between 0-33 and a high score indicates a high level of knowledge about HPV, HPV screening tests and the HPV vaccine The "Cervical Cancer and Pap-smear Test Health Belief Model Scale" will be used to understand the situations that prevent women from taking the HPV-DNA test.

SECONDARY OUTCOMES:
Having an HPV-DNA test | From the beginning of the study until the 4th month.
  The decision of women in the experimental group to have HPV-DNA testing will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Muazez Küçükkaya, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Bayrampaşa 1 nolu ASM, Istanbul, BAYRAMPAŞA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want to share the data due to the ethical principles of the research.

REFERENCES:
- [Result] Lewandowska AM, Lewandowski T, Rudzki M, Rudzki S, Laskowska B. Cancer prevention - review paper. Ann Agric Environ Med. 2021 Mar 18;28(1):11-19. doi: 10.26444/aaem/116906. Epub 2020 Mar 12. PMID 33775063
- [Result] Ghasemi M, Savabi-Esfahani M, Noroozi M, Satari M. Prediction of cervical cancer screening: application of the information-motivation-behavioral skills model. BMC Cancer. 2024 Mar 19;24(1):351. doi: 10.1186/s12885-024-12098-9. PMID 38504202
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/